CLINICAL TRIAL: NCT05741749
Title: Immediate Implant Placement in the Posterior Region Combining Sealing Socket Abutment and Peri-implant Socket Filling.A Randomized Controlled Clinical Trial
Brief Title: Immediate Implant Placement in the Posterior Region Combining Sealing Socket Abutment and Peri-implant Socket Filling.
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Head of the Department of Periodontology, oro-dental and implant surgery, Principal Investigator, Clinical Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022/19
Record Dates: First submitted 2022-05-18; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Dental Implantation
Keywords: Sealing Socket Abutment; Immediate implant; Peri implant tissue changes

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Socket Seal Abutment (Experimental)
  Interventions: Device: Socket Seal Abutment
- Conventional Healing abutment (Active Comparator)
  Interventions: Device: Socket Seal Abutment

INTERVENTIONS:
Device: Socket Seal Abutment — Customized Healing Abutment

SUMMARY:
The primary endpoint of this study is to compare the soft tissue contour changes after immediate implant placement combined to peri-implant socket filling with a sealing socket abutment (SSA) versus a standard healing abutment. The hypothesis is that the SSA better preserves the alveolar ridge profile in the cervical region compared to a conventional healing abutment. The secondary objectives aim to evaluate 3D hard tissue changes, peri-implant bone remodeling, soft tissue health, esthetic outcomes and the patients related outcome measures.

DETAILED DESCRIPTION:
Study population

Hopeless maxillary or mandibular molars with tooth anatomy and bone anchorage allowing an immediate implant procedure: apical bone height of at least 5 mm or presence of interradicular septum, socket with intact bone walls, absence a large apical periodontitis, Patients needing tooth replacement in the posterior region (molars) will be recruited from the Department of Periodontology and Oral and Implant Surgery of the University of Liège, Belgium. All the patients will meet the following inclusion criteria: good general health (ASA I/II), more than 18 years old, smoker < 10c/day, one hopeless tooth, healthy periodontal condition, the presence of at least 2 mm of keratinized gingiva, intact buccal bone wall, adequate plaque control (FMPS ≤ 25%), adequate bone quantity allowing an immediate implant procedure (apical bone height of at least 5 mm or presence of interradicular septum) and finally written consent provided. The exclusion criteria will be: auto-immune disease or immunocompromised patients, uncontrolled diabetes, use of steroids or biphosphonates, local or systemic infection (medical treatment needed prior to entrance to the study), pregnancy or breastfeeding, alcoholism or chronically drug abuse. The local exclusion criteria will be: bone availability requiring an angulated abutment, untreated local inflammation, cyst, mucosal disease or oral lesions, local irradiation therapy, oral communication with sinus after the extraction. All the patients will have to read and sign the informed consent form prior to the surgery.

Procedures

After a local anesthesia, in both groups, experienced surgeons will proceed to minimally invasive tooth extraction of the hopeless tooth. The consecutive drills for implant placement will be carried out according to the recommendation of the manufacturer while considering the future position of the crown for a screw-retained restoration and the socket anatomy. Then, implants (TLX, SLA active, Straumann Group, Basel, Switzerland) will be placed immediately in a flapless manner and an insertion torque of at least 20Ncm will be required to continue the procedure. The remaining socket will be filled with a Deproteinized Bovine Bone Mineral DBBM (Straumann Xenograft, Straumann Group, Basel, Switzerland). Once the implant placed and the socket procedure completed the patients will be allocated either to the control group or the test group. In control group, a conventional healing abutment will be placed and the remaining gap of the socket will be closed with collagen matrix (Collacone, Straumann Group, Basel, Switzerland). In the test group, an SSA will be made immediately in a chair-side manner. A Variobase (Straumann Group, Basel, Switzerland) will be placed at the implant and Teflon will be used to protect the biomaterial and implant neck. Flowable composite will be used to start shaping the form of the future SSA. On the chair-side, the finalization of the emergence profile in a tulip concave shape by additive technique will take place. Before insertion, the SSA will be polished, cleaned and disinfected in a series of ultrasonic baths (Soapy water, water and alcohol). The insertion will be made at 15 N/cm and the access hole will be obturated with teflon and Telio (Ivoclar vivadent, Schaan, Liechtenstein). A standardized parallel peri-apical radiograph using a custom-made film holder will be taken in order to record the baseline bone level. Each patient will be instructed to rinse twice daily with an aqueous solution of 0,2% Chlorhexidine (Corsodyl®, GSK, Brentford, United Kingdom) and to avoid brushing of the area until the first recall 10-12 days later. Antibiotic will be prescribed (Amoxicillin® 500mg 3x/d during 5 days) and anti-inflammatories (Ibuprofen® 600 mg) as well as additional analgesics (Paracetamol® 500 mg) will recommended according to the patient's needs. Three months after implantation, in both groups, the abutments will be removed, the osseointegration of the implants will be checked and a CAD-CAM Zirconia monolithic crown will be placed. The transmucosal design from the SSA will replicated on the final crown and in the control group the design of the crown will be determined according to the soft tissue profile.

Follow-up evaluations and data recording will be performed 7-10 days, 3 months, 6 months and 12 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Good general health (ASA I/II),
* More than 18 years old,
* Smoker < 10c/day, one hopeless tooth,
* Healthy periodontal condition,
* Presence of at least 2 mm of keratinized gingiva
* Intact buccal bone wall
* Adequate plaque control (FMPS ≤ 25%)
* Adequate bone quantity allowing an immediate implant procedure (apical bone height of at - Least 5 mm or presence of interradicular septum)
* Written consent provided

Exclusion Criteria:

* Auto-immune disease or immunocompromised patients
* Uncontrolled diabetes
* Use of steroids or biphosphonates
* Local or systemic infection (medical treatment needed prior to entrance to the study)
* Pregnancy or breastfeeding
* Alcoholism or chronically drug abuse
* Bone availability requiring an angulated abutment
* Untreated local inflammation
* Cyst
* Mucosal disease or oral lesions
* Local irradiation therapy
* Oral communication with sinus after the extraction

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change of Soft Tissue Contour from baseline to 3 months, 6 months and 1 year | 3 months, 6 months, 1 year
  Compare the soft tissue contour changes after immediate implant placement combined to peri-implant socket filling with a sealing socket abutment (SSA) versus a standard healing abutment.

SECONDARY OUTCOMES:
3D hard tissue changes | Baseline, 1 year
  Assessment of bone dimension changes
Peri-implant bone remodeling | 3 months, 6 months, 1 year
  Assessment of bone height changes
Soft tissue health changes assessed by Probing Pocket Depth | 3 months, 6 months, 1 year
  Assessed of probing depth
Soft tissue health changes assessed by Bleeding on Probing | 3 months, 6 months, 1 year
  Assessment of the bleeding percentage
Soft tissue health changes assessed by Plaque Index | 3 months, 6 months, 1 year
  Assessment of plaque percentage
Esthetic outcomes changes | 10 days, 3 months, 6 months, 12 months
  Assessed by Pink Esthetic Score (Papilla presence, tissue contour, gingival level, alveolar process, colouring and texture) as well as intra-oral photographs
Patients Related Outcome Measures | 6 months, 1 year
  Assessed by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No